CLINICAL TRIAL: NCT06675526
Title: Detour: a Smartphone Game to Help Youth Quit Smoking
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Behavioural Science Institute (Other)
Collaborators: Erasmus Medical Center (Other); Stichting Trimbos-Instituut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Detour; 12946 (Other Grant/Funding Number: KWF kankerbestrijding); KA154-YOU-000100302 (Other Grant/Funding Number: Erasmus +)
Record Dates: First submitted 2024-07-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Smoking Cessation; Smoking Reduction; Adolescent Behavior; Social Behavior
Keywords: Behaviour change; Game intervention; Peer influence; Smoking cessation; Youth
MeSH Terms: conditions — Smoking Cessation; Smoking Reduction; Adolescent Behavior; Social Behavior

STUDY DESIGN:
Intervention Model Description: A two-armed RCT (Detour vs digital self-help material to quit smoking as the control group) will be conducted to test the efficacy of Detour.
  All participants fill out Qualtrics questionnaires comprising self-report measures at screening, pre-test, post-test, 3-month follow-up, and 6-month follow-up. In addition, participants in the game group answer some questions in the mobile application, participant in-game behaviour (such as time spent playing) is measured, and text-data from the player chat room and social shell will be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Detour (Experimental): Participants have access to Detour for 5 weeks encompassing various elements: (1) Completing a stop plan during the initial week preceding the quit attempt. (2) Engaging in ecological momentary assessments, measuring affect, nicotine withdrawal, and smoking behavior during the first two weeks: one week prior to and one week post quit attempt. (3) Accessing the game for a duration of 4 weeks following the quit attempt. (4) Participating in the social shell, in which participants join private social media channels on Instagram and/or TikTok for the entirety of the intervention period.
  Interventions: Behavioral: Detour
- Digital self-help material (Active Comparator): Participants receive a self-help digital brochure, "Jouw eigen plan om te stoppen met roken" for smoking cessation in the control group. They will read this on personal demand.
  Interventions: Behavioral: Self-help brochure

INTERVENTIONS:
Behavioral: Detour — "Detour" is a mobile game designed to assist youth with smoking cessation. First, Detour targets stimuli devaluation using a gamified go/no-go training. Second, the researchers aimed to reduce delay discounting in two ways; 1) players can replace neutral images in the go/no-go training with positive images from their own lives related to their future self; 2) players can set and monitor personal goals via the game, to promote future-self priming. Third, participants join a social shell comprising Instagram and TikTok content to provide psychoeducation about quitting smoking and to interact with fellow players who quit simultaneously. Finally, the timing and content of in-game messaging is personalized to each participant based on information provided in an ecological momentary assessment component and a stop plan filled out during the week before the quit attempt.
  Arms: Detour
Behavioral: Self-help brochure — The brochure provides guidelines to independently design a stop-plan including questions about seeking support from others, strategies to fight cravings, and setting rewards for milestones after quitting. Participants will be encouraged to complete this stop-plan in week 0 of the intervention, so the week before quit day. Additionally, the brochure includes psychoeducational information that is valuable when planning to quit smoking.
  Arms: Digital self-help material

SUMMARY:
The researchers are testing a mobile game (named Detour) to support smoking cessation in adolescents and young adults (16-25 years). The game will be tested in a randomized-controlled trial (RCT) where Detour is tested against a digital self-help brochure ("Jouw eigen plan om te stoppen met roken" [in English: Your personal plan to quit smoking]) as the active control group. The researchers will recruit 604 participants (aged 16-25) and randomly assign them to receive the game or brochure intervention. The duration between pre-test and post-test for both groups is 5 weeks during which participants can access (parts of) their respective intervention. All participants quit smoking at the end of week 1 of the intervention period. Data is collected on smoking behaviour, intervention usage, and emotional well-being.

DETAILED DESCRIPTION:
The aim of the present two-armed randomized controlled trial is to test the efficacy of Detour, a smartphone game to help youth (16-25 years) quit smoking. It is designed to be an accessible, multi-component intervention providing in-the-moment distractions from cravings. First, Detour targets stimuli devaluation using a gamified go/no-go training in an endless runner game format. Second, the researchers aimed to reduce delay discounting in two ways; 1) players can replace neutral images in the go/no-go training with positive images from their own lives related to their future self; 2) players can set and monitor personal goals via the game, to promote future-self priming. Third, participants join a social shell comprising Instagram and TikTok content to provide psychoeducation about quitting smoking and to interact with fellow players who quit simultaneously. Finally, the timing and content of in-game messaging is personalized to each participant based on information provided in an ecological momentary assessment component and a stop plan filled out during the week before the quit attempt.

Detour will be tested against a self-help digital brochure, "Jouw eigen plan om te stoppen met roken" by the Trimbos Institute, the Netherlands. The brochure provides guidelines to independently design a stop-plan including questions about seeking support from others, strategies to fight cravings, and setting rewards for milestones after quitting. Additionally, the brochure has psychoeducational information that is valuable when planning to quit smoking.

For the data collection procedure, the researchers will first broadly distribute a short screening questionnaire via educational institutes and social media to assess study inclusion criteria. Eligible participants will be contacted by phone/text message/email to explain the purpose of the study further and invited to fill out the pre-test measurement if they would like to participate. The researchers will recruit nationwide and strive for a diverse sample in terms of gender, demographic location and educational levels. Participants will provide informed consent at both the screening and pre-test phases.

After the pre-test, blocks of 6 participants are randomly assigned to either the "Detour" game group or the brochure group to begin the intervention. The intervention period lasts for five weeks. During week 0 or the preparatory week, participants can access Detour or the brochure but have not yet quit. On day 1 of week 1, known as quit day, participants will quit smoking and try to remain smoke-free for the next four weeks (weeks 1-4).

The target sample size is N = 604, with 10% drop-outs taken into account. Recruitment will stop once 604 participants have received an intervention or on August 1, 2025.

The aim is to achieve 25% abstinence rates at 6-month follow-up in the game group. The researchers aim to prove a small effect size (odds ratio 1.88) with 90% power. A power analysis (logistic regression analysis, one-tailed alpha .05, and a fifty-fifty distribution of participants in both groups) showed that they will need N = 604 participants, taking into account a 10% loss.

To assess the immediate effectiveness of the game for smoking cessation in youth, logistic regression analyses will be performed with intervention group (game or brochure), as predictor and 14-day point prevalence of smoking abstinence (yes/no) at 6-month follow-up as the outcome. Age, Gender, socioeconomic status (SES), and baseline weekly smoking will be added to the model as controlled variables.

To assess the longer-term effectiveness of the game for smoking cessation in youth, logistic regression analyses will be performed with intervention group (game or brochure), as predictor and 14-day point prevalence of smoking abstinence (yes/no) at post-test as the outcome. Age, Gender, socioeconomic status (SES), and baseline weekly smoking will be added to the model as controlled variables.

To assess the effect of the game on weekly smoking, multilevel regression analysis will be performed with intervention group (game or brochure), time (pre-test, post-test, 3-month follow-up and 6-month follow-up), and their interaction as predictors, and weekly smoking as the outcome. The following models will be tested. Age, Gender, socioeconomic status (SES), and baseline weekly smoking will be added to the model as controlled variables.

* Model0 ← WeeklySmoking ~ (1 | ID); check intra-class correlations
* Model1 ← WeeklySmoking ~ TreatmentGroup + Time + Gender + Age + SES + Baseline weekly smoking + (1 | ID)
* Model2 ← WeeklySmoking~ TreatmentGroup + Time + Gender + Age + SES + Baseline weekly smoking + (1 + time | ID); compare model 1 and model 2 to see if random slopes give better model fit.
* Model3 ← WeeklySmoking~ TreatmentGroup + Time + TreatmentGroup:Time + Gender

  * Age + SES + Baseline weekly smoking + (1 + time | ID); Calculate simple slopes for both cases of treatment group.

For the analyses of the primary and secondary outcomes, a one-tailed p < .05 criteria will be used. For remaining analyses the standard p < .05 criteria will be used.

Furthermore, the intention to treat approach will be used, where it is assumed that people who missed post-test or either follow-up are non-abstinent.

Participants who only responded to the pretest but neither post-test, 3-month follow-up, nor 6-month follow-up will be considered as relapsers in analyses with abstinence as the outcome. In models with weekly smoking as the outcome, the majority of weekly smoking values would need to be imputed, so instead participants who only responded to the pre-test measure will be excluded.

The present pre-registration only pertains to the efficacy of the intervention. A follow-up registration on the in-depth analysis of the intervention effects and sub-group analyses to test who the intervention worked best for will be made. Please refer to the project page for more information (https://osf.io/k784a/).

ELIGIBILITY:
Inclusion Criteria:

1. aged 16 to 25 years
2. smokes at least weekly
3. motivated to quit smoking (participants should answer "misschien", "waarschijnlijk" or "heel erg" to the question are you motivated to quit smoking at this specific moment?).
4. installed Detour application; only applicable for participants assigned to the game intervention group.

Exclusion Criteria:

1. younger than 16 or older than 25
2. smoke less than once a week
3. not motivated to quit smoking are not eligible for this study i.e. participants who answered "helemaal niet"/"not at all") or "onwaarschijnlijk"/"unlikely" to the question are you motivated to quit smoking at this specific moment?).

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 604 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Smoking abstinence | 6 month follow-up
  The primary outcome measure will be 14-day point prevalence abstinence (yes/no) at six month follow-up i.e. 6 months from quit date.

SECONDARY OUTCOMES:
Smoking abstinence | immediate post-test after 5-week intervention period
  The primary outcome measure will be 14-day point prevalence abstinence (yes/no) at post test immediately after the 5-week intervention period.
Weekly smoking | pre-test, immediate post-test after 5-week intervention period, 3-month follow-up, and 6-month follow-up
  Weekly smoking behavior will be assessed with two questions 1) "How many days per week do you smoke on average?" and "On a day that you smoke, how many cigarettes do you smoke on average?". Weekly smoking behaviour will be assessed at pre-test within the week before the intervention begins, at immediate post-test after 5-week intervention period, at 3-month follow-up from quit date, and at 6-month follow-up from quit date. The answers to these questions will be multiplied to come to a single measure of weekly smoking. If participants remain abstinent, weekly smoking will be set to 0.

CONTACTS AND LOCATIONS:
Overall Officials: Maartje Luijten, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The researchers will share the data and analytic code in OSF and via SURFdrive, following their institute's policy.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Once the associated paper is published, anonymised data will be made openly available via the project page on OSF (https://osf.io/k784a/) with no end date.